CLINICAL TRIAL: NCT04071405
Title: Korea Post-marketing Surveillance for Xeljanz (Registered) in Ulcerative Colitis Patients
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A3921343
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Results first posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-04

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative colitis; Autoimmune Diseases; Immune System Diseases; Tofacitinib; Molecular Mechanisms of Pharmacological Action; Jak inhibitor; safety
MeSH Terms: conditions — Colitis, Ulcerative; Autoimmune Diseases; Immune System Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other

INTERVENTIONS:
Other: Non-intervention — Non-intervention observational study

SUMMARY:
As required for new medications approved by the Ministry of Food and Drug Safety, safety and efficacy information should be provided for a minimum of 90 patients treated in the setting of routine practice during 4 years following approval (until 19 September 2022). Out of all the enrolled patients, at least 18 cases (20%) will be followed up until the 52nd week to see the long term safety of Xeljanz.

DETAILED DESCRIPTION:
This is an open-label, non-comparative, non-interventional, prospective, and multi-center study conducted in Korean health care centers by accredited physicians (ie, investigators). The study population will be adult patients with moderately to severely active UC who have had an inadequate response or intolerance to the basic treatments or biological agents. Clinical Severity of Ulcerative Colitis is classified as mild, moderate, or severe based on the Mayo score or partial Mayo score. Xeljanz will be administered according to the "Dosage and Administration" of the approved labeling. There is no visit or activity mandated by this study. The investigator will collect patient data and record the information on each patient's case report form (CRF).

ELIGIBILITY:
Inclusion Criteria:

* Adult ulcerative colitis patients with moderately to severely active disease who has received at least 1 dose of Xeljanz according to the local labeling

Exclusion Criteria:

* Patients meeting any of the following criteria as per local labeling will not be included in the study.

  1. Patients with a history of hypersensitivity to any ingredients of this product.
  2. Patients with serious infection (sepsis, etc.) or active infection including localized infection.
  3. Patients with active tuberculosis.
  4. Patients with severe hepatic function disorder.
  5. Patients with an absolute neutrophil count (ANC) <1,000 cells/mm3.
  6. Patients with a lymphocyte count <500 cells/mm3.
  7. Patients with a hemoglobin level <9 g/dL.
  8. Pregnant or possibly pregnant women.
  9. Because of lactose contained in this drug, it should not be administered to patients with hereditary problems of galactose intolerance, Lapp lactase deficiency or glucose galactose malabsorption.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 19 years and older with moderately to severely active ulcerative colitis
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2020-05-12 (Actual); Primary Completion 2022-09-26 (Actual); Study Completion 2022-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Yoon H, Ye BD, Kang SB, Lee KM, Choi CH, Jo JY, Woo J, Cheon JH. Safety and effectiveness of tofacitinib in Korean adult patients with ulcerative colitis: post-marketing surveillance study. BMC Gastroenterol. 2024 Aug 19;24(1):273. doi: 10.1186/s12876-024-03336-2. PMID 39160459
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A3921343

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult participants with moderately to severely active ulcerative colitis (UC) who had an inadequate response or intolerance to basic treatments or biological agents and were prescribed Xeljanz (tofacitinib) for the first time as part of routine practice at Korean healthcare centers were observed in this post-marketing surveillance study.
Groups:
- Tofacitinib: Participants with moderately to severely active ulcerative colitis who had an inadequate response or intolerance to basic treatments or biological agents and received tofacitinib as part of routine practice at Korean health care centers were observed.
Period: Overall Study
Arm/Group | Tofacitinib
Started | 110
Safety Population | 107
Completed | 107
Not Completed | 3
Not completed — Protocol Violation | 3

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants registered for this study who were prescribed at least 1 dose of Xeljanz according to the local label and followed up for safety data.
Arm/Group | Tofacitinib
Number analyzed (Participants) | 107
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.83 (13.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 76
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events, Adverse Drug Reactions, Serious Adverse Events and Serious Adverse Drug Reactions
Description: An adverse event (AE) was any untoward medical occurrence in a participant administered a medicinal product which need not necessarily have causal relationship with product treatment or usage. Serious adverse event was any adverse event that resulted in any of the following outcomes or deemed significant for any other reason: death; life-threatening; initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly. Adverse drug reaction (ADR) was any untoward medical occurrence attributed to Xeljanz. Serious ADR: any ADR resulting in any of following outcomes or deemed significant for any other reason: death; life-threatening; initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly. 95% confidence interval (CI) was based on Clopper-Pearson method. This outcome measure is reported for all participants including long term users (i.e. treated with Xeljanz for at least 52 weeks).
Time Frame: From first dose of Xeljanz until 52 weeks
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 107
Percentage of participants
  Adverse events | 40.19 [30.82 to 50.11]
  Adverse drug reactions | 24.30 [16.53 to 33.54]
  Serious adverse events | 7.48 [3.28 to 14.20]
  Serious adverse drug reactions | 0.93 [0.02 to 5.10]

2. Primary Outcome: Number of Participants With Adverse Events, Adverse Drug Reactions, Serious Adverse Events and Serious Adverse Drug Reactions in Long Term Users
Description: An adverse event (AE) was any untoward medical occurrence in a participant administered a medicinal product which need not necessarily have causal relationship with product treatment or usage. A serious adverse event was any adverse event that resulted in any of the following outcomes or deemed significant for any other reason: death; life-threatening; initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly. An adverse drug reaction (ADR) was any untoward medical occurrence attributed to Xeljanz. Serious ADR: any ADR resulting in any of following outcomes or deemed significant for any other reason: death; life-threatening; initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly. This outcome measure was analyzed only in long term users.
Time Frame: From first dose of Xeljanz until 52 weeks
Population: Safety analysis set included all participants registered for this study who were prescribed at least 1 dose of Xeljanz according to the local label and followed up for safety data. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 60
Participants
  Adverse events | 27
  Adverse drug reactions | 18
  Serious adverse events | 3
  Serious adverse drug reactions | 0

3. Primary Outcome: Percentage of Participants With Unexpected Adverse Events (AE), Unexpected Adverse Drug Reactions, Unexpected Serious Adverse Events (SAE), and Unexpected Serious Adverse Drug Reactions
Description: Unexpected AE: any event that may be symptomatically, pathophysiologically related to event listed in labeling, but differed from labeled event because of greater severity or specificity. ADR: any untoward medical occurrence attributed to Xeljanz. All events that were not included in "Precautions for use" section of local product document were classified as "unexpected" adverse drug reactions. Serious ADR: any ADR resulting in any of following outcomes or deemed significant for any other reason: death; life-threatening; initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly. SAE: any untoward medical occurrence in participant administered medicinal/nutritional product at any dose that resulted in death was life-threatening. 95% CI was based on Clopper-Pearson method. This outcome measure is reported for all participants including long term users.
Time Frame: From first dose of Xeljanz until 52 weeks
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 107
Percentage of participants
  Unexpected adverse events | 22.43 [14.93 to 31.51]
  Unexpected adverse drug reactions | 12.15 [6.63 to 19.88]
  Unexpected serious adverse events | 3.74 [1.03 to 9.30]
  Unexpected serious adverse drug reactions | 0 [0 to 0]

4. Primary Outcome: Number of Participants With Unexpected Adverse Events, Unexpected Adverse Drug Reactions, Unexpected Serious Adverse Events, and Unexpected Serious Adverse Drug Reactions in Long Term Users
Description: Unexpected AE: any event that may be symptomatically, pathophysiologically related to event listed in labeling, but differed from labeled event because of greater severity or specificity. ADR: any untoward medical occurrence attributed to Xeljanz. All events that were not included in "Precautions for use" section of local product document were classified as "unexpected" adverse drug reactions. Serious ADR: any ADR resulting in any of following outcomes or deemed significant for any other reason: death; life-threatening; initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly. SAE: any untoward medical occurrence in participant administered medicinal/nutritional product at any dose that resulted in death was life-threatening. This outcome measure was analyzed only in long term users.
Time Frame: From first dose of Xeljanz until 52 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 60
Participants
  Unexpected adverse events | 13
  Unexpected adverse drug reactions | 9
  Unexpected serious adverse events | 1
  Unexpected serious adverse drug reactions | 0

5. Primary Outcome: Percentage of Participants With Adverse Events of Special Interest
Description: An adverse event was any untoward medical occurrence in a participant administered a medicinal product. The event need not necessarily have a causal relationship with the product treatment or usage. Adverse events of special interest were defined as serious or non-serious AEs which were of scientific and medical concern specific to the investigational product. 95% CI was based on Clopper-Pearson method. This outcome measure is reported for all participants including long term users.
Time Frame: From first dose of Xeljanz until 52 weeks
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 107
Percentage of participants | 1.87 [0.23 to 6.59]

6. Primary Outcome: Number of Participants With Adverse Events of Special Interest in Long Term Users
Description: An adverse event was any untoward medical occurrence in a participant administered a medicinal product. The event need not necessarily have a causal relationship with the product treatment or usage. Adverse events of special interest were defined as serious or non-serious AEs which were of scientific and medical concern specific to the investigational product. This outcome measure was analyzed only in long term users.
Time Frame: From first dose of Xeljanz until 52 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 60
Participants | 2

7. Primary Outcome: Number of Participants With Adverse Events by Their Severity
Description: An adverse event was any untoward medical occurrence in a participant administered a medicinal product. The event need not necessarily have a causal relationship with the product treatment or usage. AEs were categorized as per the severity: mild: did not cause any significant problem to the participant, administration of medicinal product continued without dose adjustment; moderate: caused a problem that did not interfere significantly with usual activities or the clinical status, dose of the medicinal product was adjusted or other therapy was added due to the AE; severe: caused a problem that interfered significantly with usual activities, or the clinical status and the medicinal product was stopped due to AE. One participant may experience more than one event; hence, one participant may be included in more than one category specified below. This outcome measure is reported for all participants including long term users.
Time Frame: From first dose of Xeljanz until 52 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 43
Participants
  Mild | 35
  Moderate | 11
  Severe | 4

8. Primary Outcome: Number of Participants With Adverse Events by Their Severity in Long Term Users
Description: An adverse event was any untoward medical occurrence in a participant administered a medicinal product. The event need not necessarily have a causal relationship with the product treatment or usage. AEs were categorized as per the severity: mild: did not cause any significant problem to the participant, administration of medicinal product continued without dose adjustment; moderate: caused a problem that did not interfere significantly with usual activities or the clinical status, dose of the medicinal product was adjusted or other therapy was added due to the AE; severe: caused a problem that interfered significantly with usual activities, or the clinical status and the medicinal product was stopped due to AE. One participant may experience more than one event; hence, one participant may be included in more than one category specified below. This outcome measure was analyzed only in long term users.
Time Frame: From first dose of Xeljanz until 52 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 27
Participants
  Mild | 24
  Moderate | 4
  Severe | 1

9. Primary Outcome: Number of Participants With Adverse Events by Their Outcomes
Description: An AE was any untoward medical occurrence in a participant administered a medicinal product. The event need not necessarily have a causal relationship with the product treatment or usage. AE outcomes were categorized as: recovered; recovered with sequelae; recovering; not recovered; unknown. One participant may experience more than one event; hence, one participant may be included in more than one category specified below. This outcome measure is reported for all participants including long term users.
Time Frame: From first dose of Xeljanz until 52 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 43
Participants
  Recovered | 33
  Recovered with sequelae | 0
  Recovering | 13
  Not recovered | 6
  Unknown | 1

10. Primary Outcome: Number of Participants With Adverse Events by Their Outcomes in Long Term Users
Description: An AE was any untoward medical occurrence in a participant administered a medicinal product. The event need not necessarily have a causal relationship with the product treatment or usage. AE outcomes were categorized as: recovered; recovered with sequelae; recovering; not recovered; unknown. One participant may experience more than one event; hence, one participant may be included in more than one category specified below. This outcome measure was analyzed only in long term users.
Time Frame: From first dose of Xeljanz until 52 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 27
Participants
  Recovered | 21
  Recovered with sequelae | 0
  Recovering | 7
  Not recovered | 3
  Unknown | 1

11. Primary Outcome: Number of Participants With Adverse Events by Their Seriousness
Description: An adverse event was any untoward medical occurrence in a participant administered a medicinal product. The event need not necessarily have a causal relationship with the product treatment or usage. Adverse events were classified as per their seriousness as following: results in death, is life-threatening, requires inpatient hospitalization or prolongation of hospitalization, results in persistent or significant disability/incapacity, results in congenital anomaly/birth defect, other important medical event. One participant may experience more than one event; hence, one participant may be included in more than one category specified below. This outcome measure is reported for all participants including long term users.
Time Frame: From first dose of Xeljanz until 52 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 43
Participants
  Results in death | 0
  Life-threatening | 0
  Requires inpatient hospitalization or prolongation of hospitalization | 8
  Results in persistent or significant disability/incapacity | 0
  Results in congenital anomaly/birth defect | 0
  Other important medical event | 0
  Non-Serious | 41

12. Primary Outcome: Number of Participants With Adverse Events by Their Seriousness in Long Term Users
Description: An adverse event was any untoward medical occurrence in a participant administered a medicinal product. The event need not necessarily have a causal relationship with the product treatment or usage. Adverse events were classified as per their seriousness as following: results in death, was life-threatening, required inpatient hospitalization or prolongation of hospitalization, resulted in persistent or significant disability/incapacity, results in congenital anomaly/birth defect, other important medical event. One participant may experience more than one event; hence, one participant may be included in more than one category specified below. This outcome measure was analyzed only in long term users.
Time Frame: From first dose of Xeljanz until 52 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 27
Participants
  Results in death | 0
  Is life-threatening | 0
  Requires inpatient hospitalization or prolongation of hospitalization. | 3
  Results in persistent or significant disability/incapacity | 0
  Results in congenital anomaly/birth defect | 0
  Other important medical event | 0
  Non-Serious | 26

13. Primary Outcome: Number of Participants With Adverse Events by Action Taken
Description: An adverse event was any untoward medical occurrence in a participant administered a medicinal product. The event need not necessarily have a causal relationship with the product treatment or usage. Action taken with regard to the medicinal product included: permanently discontinued; temporarily discontinued or delayed; dose reduced; dose increased; no change; and not applicable. One participant may experience more than one event; hence, one participant may be included in more than one category specified below. This outcome measure is reported for all participants including long term users.
Time Frame: From first dose of Xeljanz until 52 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 43
Participants
  Permanently discontinued | 8
  Temporary discontinued or delayed | 2
  Dose reduced | 2
  Dose increased | 3
  No change | 35
  Not applicable | 1

14. Primary Outcome: Number of Participants With Adverse Events by Action Taken in Long Term Users
Description: An adverse event was any untoward medical occurrence in a participant administered a medicinal product. The event need not necessarily have a causal relationship with the product treatment or usage. Action taken with regard to the medicinal product included: permanently discontinued; temporarily discontinued or delayed; dose reduced; dose increased; no change; and not applicable. One participant may experience more than one event; hence, one participant may be included in more than one category specified below. This outcome measure was analyzed only in long term users.
Time Frame: From first dose of Xeljanz until 52 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 27
Participants
  Permanently discontinued | 0
  Temporary discontinued or delayed | 0
  Dose reduced | 1
  Dose increased | 2
  No change | 26
  Not applicable | 0

15. Primary Outcome: Number of Participants With Adverse Events by Their Causality Assessment
Description: An AE was any untoward medical occurrence in a participant when administered a medicinal product. The event need not necessarily have a causal relationship with the product treatment or usage. Causal relationship of AEs to the medicinal product was allocated by the investigator according to the following criteria: certain, probable/likely, possible, unlikely, conditional/unclassified, unassessible/unclassifiable, not applicable. One participant may experience more than one event; hence, one participant may be included in more than one category specified below. This outcome measure is reported for all participants including long term users.
Time Frame: From first dose of Xeljanz until 52 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 43
Participants
  Certain | 1
  Probable/likely | 0
  Possible | 9
  Unlikely | 22
  Conditional/ unclassified | 6
  Unassessible/ unclassifiable | 13
  Not applicable | 0

16. Primary Outcome: Number of Participants With Adverse Events by Their Causality Assessment in Long Term Users
Description: An AE was any untoward medical occurrence in a participant when administered a medicinal product. The event need not necessarily have a causal relationship with the product treatment or usage. Causal relationship of AEs to the medicinal product was allocated by the investigator according to the following criteria: certain, probable/likely, possible, unlikely, conditional/unclassified, unassessible/unclassifiable, not applicable. One participant may experience more than one event; hence, one participant may be included in more than one category specified below. This outcome measure was analyzed only in long term users.
Time Frame: From first dose of Xeljanz until 52 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 27
Participants
  Certain | 0
  Probable/likely | 0
  Possible | 4
  Unlikely | 11
  Conditional/unclassified | 5
  Unassessible/unclassifiable | 11
  Not applicable | 0

17. Primary Outcome: Number of Participants With Adverse Events by Their Other Causality Assessment
Description: An AE was any untoward medical occurrence in a participant when administered a medicinal product. The event need not necessarily have a causal relationship with the product treatment or usage. Adverse events by their other causality assessment (in case of unlikely) were classified as: Disease under the study, Other diseases, Concomitant treatment medication or non-medication, and Other. One participant may experience more than one event; hence, one participant may be included in more than one category specified below. This outcome measure is reported for all participants including long term users.
Time Frame: From first dose of Xeljanz until 52 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 22
Participants
  Disease under the study | 13
  Other diseases | 5
  Concomitant treatment medication or non-medication | 2
  Other | 5

18. Primary Outcome: Number of Participants With Adverse Events by Their Other Causality Assessment in Long Term Users
Description: An AE was any untoward medical occurrence in a participant when administered a medicinal product. The event need not necessarily have a causal relationship with the product treatment or usage. Adverse events by their other causality assessment (in case of unlikely) were classified as: Disease under the study, Other diseases, Concomitant treatment medication or non-medication, and Other. One participant may experience more than one event; hence, one participant may be included in more than one category specified below. This outcome measure included only long term users. This outcome measure was analyzed only in long term users.
Time Frame: From first dose of Xeljanz until 52 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 11
Participants
  Disease under the study | 6
  Other diseases | 3
  Concomitant treatment medication or non-medication | 1
  Other | 2

19. Secondary Outcome: Mayo Index, Mayo Score and Partial Mayo Score at Baseline, Week 8, Week 16 and Week 24
Description: Mayo score (MS): measured disease activity (DA) of UC; total score range=0 to 12, higher score=severe DA. Mayo index was based on 4 clinical evaluation criteria: Stool frequency, Rectal bleeding, Endoscopy finding, Physician's global assessment(PGA).Each sub-score range=0 to 3,higher score=more severe DA.Stool frequency:0=normal number of stool, 1=1 to 2 stool/day >normal, 2=3 to 4 stool/day >normal, 3= >4 stool/day >normal; Rectal bleeding:0=None,1=Visible blood with stool less than half time, 2=Visible blood with stool>half time, 3=Mostly blood with rare stool; Endoscopic finding:0=Normal/inactive, 1=Mild with erythema, decreased vascular pattern, mild friability, 2=Moderate with marked erythema, absent vascular pattern, friability, erosion, 3=Severe with spontaneous bleeding, ulceration, pseudopolyp; PGA: 0=Normal/inactive, 1=Mild, 2=Moderate, 3=severe Partial MS=sum of all evaluation criteria, except endoscopy finding.Partial MS score range=0 to 9;higher score=more severe DA.
Time Frame: Baseline, Week 8, Week 16 and Week 24
Population: Effectiveness analysis included all participants who had participated in safety analysis, whose effectiveness data available after 24 weeks of treatment or based on the last assessment performed at the time of treatment discontinuation if participant did not complete the 24 weeks of treatment. If. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure. 'Number Analyzed (n)' signifies participants evaluable for specified rows.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib
Number analyzed (Participants) | 101
Units on a scale
  Stool frequency (Baseline) | 2.41 (0.70)
  Rectal bleeding (Baseline) | 1.57 (0.84)
  Physician's global assessment (Baseline) | 2.15 (0.62)
  Finding of endoscopy (Baseline): number analyzed (Participants) | 98
  Finding of endoscopy (Baseline) | 2.56 (0.56)
  Mayo score (Baseline): number analyzed (Participants) | 98
  Mayo score (Baseline) | 8.64 (1.56)
  Partial Mayo score (Baseline) | 6.13 (1.40)
  Stool frequency (Week 8): number analyzed (Participants) | 87
  Stool frequency (Week 8) | 1.23 (1.12)
  Rectal bleeding (Week 8): number analyzed (Participants) | 87
  Rectal bleeding (Week 8) | 0.53 (0.74)
  Physician's global assessment (Week 8): number analyzed (Participants) | 87
  Physician's global assessment (Week 8) | 0.82 (0.87)
  Finding of endoscopy (Week 8): number analyzed (Participants) | 7
  Finding of endoscopy (Week 8) | 1.14 (1.07)
  Mayo score (Week 8): number analyzed (Participants) | 7
  Mayo score (Week 8) | 4.00 (3.56)
  Partial Mayo score (Week 8): number analyzed (Participants) | 87
  Partial Mayo score (Week 8) | 2.57 (2.28)
  Stool frequency (Week 16): number analyzed (Participants) | 91
  Stool frequency (Week 16) | 0.86 (0.96)
  Rectal bleeding (Week 16): number analyzed (Participants) | 91
  Rectal bleeding (Week 16) | 0.30 (0.57)
  Physician's global assessment (Week 16): number analyzed (Participants) | 91
  Physician's global assessment (Week 16) | 0.60 (0.74)
  Finding of endoscopy (Week 16): number analyzed (Participants) | 64
  Finding of endoscopy (Week 16) | 1.44 (1.08)
  Mayo score (Week 16): number analyzed (Participants) | 64
  Mayo score (Week 16) | 3.17 (2.67)
  Partial Mayo score (Week 16): number analyzed (Participants) | 91
  Partial Mayo score (Week 16) | 1.76 (1.91)
  Stool frequency (Week 24): number analyzed (Participants) | 60
  Stool frequency (Week 24) | 0.80 (0.92)
  Rectal bleeding (Week 24): number analyzed (Participants) | 60
  Rectal bleeding (Week 24) | 0.30 (0.56)
  Physician's global assessment (Week 24): number analyzed (Participants) | 60
  Physician's global assessment (Week 24) | 0.42 (0.59)
  Finding of endoscopy (Week 24): number analyzed (Participants) | 2
  Finding of endoscopy (Week 24) | 0.50 (0.71)
  Mayo score (Week 24): number analyzed (Participants) | 2
  Mayo score (Week 24) | 1.00 (1.41)
  Partial Mayo score (Week 24): number analyzed (Participants) | 60
  Partial Mayo score (Week 24) | 1.52 (1.71)

20. Secondary Outcome: Mayo Index, Mayo Score and Partial Mayo Score at Week 8, Week 16, Week 24 and Week 52 for Long Term Users
Description: Mayo score (MS): measured disease activity (DA) of UC; total score range=0 to 12, higher score=severe DA. Mayo index was based on 4 clinical evaluation criteria: Stool frequency, Rectal bleeding, Endoscopy finding, Physician's global assessment (PGA). Each sub-score range=0 to 3,higher score=more severe DA. Stool frequency:0=normal number of stool, 1=1 to 2 stool/day >normal, 2=3 to 4 stool/day >normal, 3= >4 stool/day >normal; Rectal bleeding:0=None,1=Visible blood with stool less than half time, 2=Visible blood with stool>half time, 3=Mostly blood with rare stool; Endoscopic finding:0=Normal/inactive, 1=Mild with erythema, decreased vascular pattern, mild friability, 2=Moderate with marked erythema, absent vascular pattern, friability, erosion, 3=Severe with spontaneous bleeding, ulceration, pseudopolyp; PGA: 0=Normal/inactive, 1=Mild, 2=Moderate, 3=severe. Partial MS=sum of all evaluation criteria, except endoscopy finding.Partial MS score range=0 to 9; higher score=more severe DA.
Time Frame: Baseline, Week 8, Week 16, Week 24 and Week 52
Population: Effectiveness analysis included all participants who had participated in safety analysis, whose effectiveness data available after 24 weeks of treatment. Here, 'Overall Number of participants Analyzed' signifies participants evaluable for this outcome measure. 'Number Analyzed' signifies participants evaluable for specified rows.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib
Number analyzed (Participants) | 60
Units on a scale
  Stool frequency (Baseline) | 2.38 (0.72)
  Rectal bleeding (Baseline) | 1.48 (0.91)
  Physician's global assessment (Baseline) | 2.08 (0.65)
  Finding of endoscopy (Baseline) | 2.55 (0.57)
  Mayo score (Baseline) | 8.5 (1.55)
  Partial score (Baseline) | 5.95 (1.42)
  Stool frequency (Week 8): number analyzed (Participants) | 49
  Stool frequency (Week 8) | 0.96 (1.04)
  Rectal bleeding (Week 8): number analyzed (Participants) | 49
  Rectal bleeding (Week 8) | 0.43 (0.71)
  Physician's global assessment (Week 8): number analyzed (Participants) | 49
  Physician's global assessment (Week 8) | 0.65 (0.75)
  Finding of endoscopy (Week 8): number analyzed (Participants) | 2
  Finding of endoscopy (Week 8) | 1.00 (0.00)
  Mayo score (Week 8): number analyzed (Participants) | 2
  Mayo score (Week 8) | 3.50 (0.71)
  Partial Mayo score (Week 8): number analyzed (Participants) | 49
  Partial Mayo score (Week 8) | 2.04 (2.02)
  Stool frequency (Week 16): number analyzed (Participants) | 59
  Stool frequency (Week 16) | 0.59 (0.72)
  Rectal bleeding (Week 16): number analyzed (Participants) | 59
  Rectal bleeding (Week 16) | 0.22 (0.46)
  Physician's global assessment (Week 16): number analyzed (Participants) | 59
  Physician's global assessment (Week 16) | 0.47 (0.60)
  Finding of endoscopy (Week 16): number analyzed (Participants) | 41
  Finding of endoscopy (Week 16) | 1.29 (1.05)
  Mayo score (Week 16): number analyzed (Participants) | 41
  Mayo score (Week 16) | 2.37 (1.88)
  Partial Mayo score (Week 16): number analyzed (Participants) | 59
  Partial Mayo score (Week 16) | 1.29 (1.44)
  Stool frequency (Week 24): number analyzed (Participants) | 47
  Stool frequency (Week 24) | 0.70 (0.81)
  Rectal bleeding (Week 24): number analyzed (Participants) | 47
  Rectal bleeding (Week 24) | 0.23 (0.48)
  Physician's global assessment (Week 24): number analyzed (Participants) | 47
  Physician's global assessment (Week 24) | 0.38 (0.57)
  Finding of endoscopy (Week 24): number analyzed (Participants) | 1
  Finding of endoscopy (Week 24) | 1.00 (NA) — Standard deviation could not be calculated for a single participant.
  Mayo score (Week 24): number analyzed (Participants) | 1
  Mayo score (Week 24) | 2.00 (NA) — Standard deviation could not be calculated for a single participant.
  Partial Mayo score (Week 24): number analyzed (Participants) | 47
  Partial Mayo score (Week 24) | 1.32 (1.52)
  Stool frequency (Week 52): number analyzed (Participants) | 50
  Stool frequency (Week 52) | 0.74 (0.85)
  Rectal bleeding (Week 52): number analyzed (Participants) | 50
  Rectal bleeding (Week 52) | 0.18 (0.44)
  Physician's global assessment (Week 52): number analyzed (Participants) | 50
  Physician's global assessment (Week 52) | 0.56 (0.67)
  Finding of endoscopy (Week 52): number analyzed (Participants) | 13
  Finding of endoscopy (Week 52) | 1.46 (1.33)
  Mayo score (Week 52): number analyzed (Participants) | 13
  Mayo score (Week 52) | 3.54 (3.48)
  Partial Mayo score (Week 52): number analyzed (Participants) | 50
  Partial Mayo score (Week 52) | 1.48 (1.57)

21. Secondary Outcome: Number of Participants With Mucosal Healing at Week 8, Week 16 and Week 24
Description: Mucosal healing was defined by Mayo or partial Mayo endoscopic score of 0 or 1 where 0=Normal/inactive disease,1=Mild disease with erythema, decreased vascular pattern, mild friability.
Time Frame: Week 8, Week 16 and Week 24
Population: Effectiveness analysis:all participants who participated in safety analysis, effectiveness data was available after 24 week(W) of treatment/based on last assessment at time of discontinuation if participant did not complete 24 W of treatment. "Overall Number of Participants Analyzed":participant evaluable for outcome measure. Participant in 'Overall Number of Participants Analyzed' contributed data to table, may not have evaluable data for each row. 'n': participant evaluable for specified row.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 73
Participants
  Week 8: number analyzed (Participants) | 7
  Week 8: Achieved | 5
  Week 8: Not achieved | 2
  Week 16: number analyzed (Participants) | 64
  Week 16: Achieved | 37
  Week 16: Not achieved | 27
  Week 24: number analyzed (Participants) | 2
  Week 24: Achieved | 2
  Week 24: Not achieved | 0

22. Secondary Outcome: Number of Participants With Mucosal Healing at Week 8, Week 16, Week 24 and Week 52 for Long Term Users
Description: as for outcome 21
Time Frame: Week 8, Week 16, Week 24 and Week 52
Population: Effectiveness analysis set: all participants who had participated in safety analysis, whose effectiveness data available after 24 weeks of treatment. "Overall Number of Participants Analyzed": participants evaluable for this outcome measure. All participants reported under 'Overall Number of Participants Analyzed' contributed data to table but may not have evaluable data for every row. 'Number Analyzed' signifies participants evaluable for specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 57
Participants
  Week 8: number analyzed (Participants) | 2
  Week 8: Achieved | 2
  Week 8: Not achieved | 0
  Week 16: number analyzed (Participants) | 41
  Week 16: Achieved | 25
  Week 16: Not achieved | 16
  Week 24: number analyzed (Participants) | 1
  Week 24: Achieved | 1
  Week 24: Not achieved | 0
  Week 52: number analyzed (Participants) | 13
  Week 52: Achieved | 6
  Week 52: Not achieved | 7

23. Secondary Outcome: Number of Participants With Remission at Week 8, Week 16 and Week 24
Description: Clinical remission was defined as Mayo score being less than or equal to 2 or partial MS <=1 and other sub-scores not more than 1. Total MS score range=0-12, where higher score=severe DA. MS based on 4 clinical evaluation criteria: Stool frequency, Rectal bleeding (RB), Finding of endoscopy, PGA. Each sub score range=0 to 3,higher score=more severe DA. Partial MS= sum of all evaluation criteria, except endoscopy finding. Partial MS total score=0 to 9 where, higher score=more severe disease activity.
Time Frame: Week 8, Week 16, and Week 24
Population: Effectiveness analysis: all participants who participated in safety analysis, effectiveness data was available after 24 week(W) of treatment/based on last assessment at time of discontinuation if participant did not complete 24 W of treatment. "Overall Number of Participants Analyzed": participant evaluable for outcome measure. Participant in 'Overall Number of Participants Analyzed' contributed data to table, may not had evaluable data for each row. 'n': participant evaluable for specified row.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 101
Participants
  Week 8: number analyzed (Participants) | 86
  Week 8: Achieved | 34
  Week 8: Not achieved | 52
  Week 16: number analyzed (Participants) | 91
  Week 16: Achieved | 42
  Week 16: Not achieved | 49
  Week 24: number analyzed (Participants) | 60
  Week 24: Achieved | 34
  Week 24: Not achieved | 26

24. Secondary Outcome: Number of Participants With Remission at Week 8, Week 16, Week 24 and Week 52 for Long Term Users
Description: as for outcome 23
Time Frame: Week 8, Week 16, Week 24 and Week 52
Population: Effectiveness analysis set: all participants who had participated in safety analysis, whose effectiveness data available after 24 weeks of treatment. Overall Number of Participants Analyzed": participants evaluable for this outcome measure. All participants reported under 'Overall Number of Participants Analyzed' contributed data to table but may not have evaluable data for every row. 'Number Analyzed' signifies participants evaluable for specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 60
Participants
  Week 8: number analyzed (Participants) | 48
  Week 8: Achieved | 23
  Week 8: Not achieved | 25
  Week 16: number analyzed (Participants) | 59
  Week 16: Achieved | 31
  Week 16: Not achieved | 28
  Week 24: number analyzed (Participants) | 47
  Week 24: Achieved | 29
  Week 24: Not achieved | 18
  Week 52: number analyzed (Participants) | 50
  Week 52: Achieved | 27
  Week 52: Not achieved | 23

25. Secondary Outcome: Number of Participants With Clinical Response at Week 8, Week 16 and Week 24
Description: Clinical response was defined as Mayo score being greater than or equal to 3 point, 30% from baseline, decrease of 1 or more in Rectal bleeding score or rectal bleeding score of 0 or 1. Total MS score range=0-12, where higher score=severe DA. MS based on 4 clinical evaluation criteria: Stool frequency, Rectal bleeding (RB), Finding of endoscopy, PGA. Each sub score range=0 to 3,higher score=more severe DA. Partial MS= sum of all evaluation criteria, except endoscopy finding. Partial MS total score=0 to 9 where, higher score=more severe disease activity.
Time Frame: Week 8, Week 16 and Week 24
Population: Effectiveness analysis: all participants who participated in safety analysis, effectiveness data was available after 24 week(W) of treatment/based on last assessment at time of discontinuation if participant did not complete 24 W of treatment."Overall Number of Participants Analyzed": participant evaluable for outcome measure.Participant under 'Overall Number of Participants Analyzed' contributed data to table,may not had evaluable data for each row.'n': participants evaluable for specified row.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 101
Participants
  Week 8: number analyzed (Participants) | 100
  Week 8: Achieved | 78
  Week 8: Not achieved | 22
  Week 16: number analyzed (Participants) | 100
  Week 16: Achieved | 88
  Week 16: Not achieved | 12
  Week 24: number analyzed (Participants) | 100
  Week 24: Achieved | 57
  Week 24: Not achieved | 43

26. Secondary Outcome: Number of Participants With Clinical Response at Week 8, Week 16, Week 24 and Week 52 for Long Term Users
Description: as for outcome 25
Time Frame: Week 8, Week 16, Week 24 and Week 52
Population: Effectiveness analysis set: all participants who had participated in safety analysis, whose effectiveness data available after 24 weeks of treatment. Here, 'Overall Number of participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 60
Participants
  Week 8: Achieved | 45
  Week 8: Not achieved | 15
  Week 16: Achieved | 58
  Week 16: Not achieved | 2
  Week 24: Achieved | 46
  Week 24: Not achieved | 14
  Week 52: Achieved | 49
  Week 52: Not achieved | 11

27. Secondary Outcome: Number of Participants According to Final Effectiveness Evaluation by Investigator
Description: The final effectiveness evaluation was determined by the investigator into 4 categories ('Improved', 'Unchanged', 'Aggravated', 'Not assessible'). Improved: Symptoms of ulcerative colitis have improved or showed adequate maintenance effect after taking Xeljanz; Unchanged: Symptoms have not changed much since taking Xeljanz; Aggravated: Symptoms have worsened after taking Xeljanz; Not assessible.
Time Frame: From first dose of Xeljanz until 24 weeks
Population: Effectiveness analysis set: all participants who had participated in safety analysis, whose effectiveness data available after 24 weeks of treatment or based on last assessment performed at time of treatment discontinuation if participant did not complete 24 weeks of treatment. Here, 'Overall Number of participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 101
Participants
  Effective, Improved | 90
  Not-effective, Unchanged | 9
  Not-effective, Aggravated | 2
  Not assessible | 0

ADVERSE EVENTS:
Time Frame: From first dose of Xeljanz until 52 weeks
Description: An AE term may be reported as both a serious and non-serious AE but are distinct events. An AE may be serious for 1 participant and non-serious for another participant, or a participant may have experienced both a serious and non-serious episode of the same event. Safety population defined as records from all participants collected into the study were included. Events were recorded from participants' clinical practice hospital documents.
Arm/Group | Tofacitinib
All-Cause Mortality (participants affected / at risk) | 0/107
Serious Adverse Events (participants affected / at risk) | 8/107
Other Adverse Events (participants affected / at risk) | 41/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tofacitinib (N=107)
Abdominal pain (Gastrointestinal disorders) | 1
Colitis ulcerative (Gastrointestinal disorders) | 2
Pouchitis (Gastrointestinal disorders) | 1
Drug ineffective (General disorders) | 1
Anal abscess (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 1
Cytomegalovirus colitis (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tofacitinib (N=107)
Anaemia (Blood and lymphatic system disorders) | 7
Abdominal pain (Gastrointestinal disorders) | 1
Colitis ulcerative (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Gastritis erosive (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Proctalgia (Gastrointestinal disorders) | 1
Chest discomfort (General disorders) | 1
Drug ineffective (General disorders) | 1
Loss of therapeutic response (General disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 3
Anal abscess (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 1
Clostridium difficile infection (Infections and infestations) | 1
Cytomegalovirus colitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Periodontitis (Infections and infestations) | 1
Spinal column injury (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 2
Blood cholesterol increased (Investigations) | 2
Blood creatinine increased (Investigations) | 1
Transaminases increased (Investigations) | 1
Vitamin D decreased (Investigations) | 1
Weight increased (Investigations) | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Increased appetite (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Essential thrombocythaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 3
Hypoaesthesia (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Amenorrhoea (Reproductive system and breast disorders) | 1
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 1
Cervical polyp (Reproductive system and breast disorders) | 1
Cervix inflammation (Reproductive system and breast disorders) | 1
Endometriosis (Reproductive system and breast disorders) | 1
Menstruation irregular (Reproductive system and breast disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
Onycholysis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-03-25): https://cdn.clinicaltrials.gov/large-docs/05/NCT04071405/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-02): https://cdn.clinicaltrials.gov/large-docs/05/NCT04071405/SAP_001.pdf